CLINICAL TRIAL: NCT00000281
Title: Pharmacotherapy for Schizophrenic Drug Users
Brief Title: Pharmacotherapy for Schizophrenic Drug Users - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-09250-6; P50DA009250 (NIH); P50-09250-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders; Shcizophrenia
Keywords: anti psychotic agents
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Amantadine

INTERVENTIONS:
Behavioral: Amantadine

SUMMARY:
The purpose of this study is to evaluate maintenance neuroleptics for Schizophrenic patients who are cocaine abusers.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-09; Primary Completion 1999-08 (Actual); Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Drug use
Retention
Psychological symptoms
Schizophrenic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Kosten, M.D., Principal Investigator — VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healthcare System, New Haven, Connecticut, United States